CLINICAL TRIAL: NCT05245838
Title: A Phase 1 Randomized, Subject-Blinded, Active-Controlled, Dose Escalation, Multicenter Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an Investigational Herpes Zoster Vaccine (Z-1018) Compared to Shingrix® in Healthy Adult Volunteers Between the Ages of 50 and 69 Years
Brief Title: Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an Investigational Herpes Zoster Vaccine (Z-1018) Compared to Shingrix® in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: DV2-ZOS-01
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Shingles; Herpes Zoster; Vaccine-Preventable Diseases
MeSH Terms: conditions — Herpes Zoster; Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Z-1018 Dose Level 1 (Experimental): 100 mcg gE + 3000 mcg CpG 1018
  Interventions: Biological: Z-1018
- Z-1018 Dose Level 1a (Experimental): 100 mcg gE + 3000 mcg CpG 1018 + alum
  Interventions: Biological: Z-1018
- Z-1018 Dose Level 2 (Experimental): 100 mcg gE + 6000 mcg CpG 1018
  Interventions: Biological: Z-1018
- Z-1018 Dose Level 2a (Experimental): 100 mcg gE + 6000 mcg CpG 1018 + alum
  Interventions: Biological: Z-1018
- Shingrix (Active Comparator)
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Z-1018 — contains gE at a dose of 100 mcg to be combined with a Toll-like receptor 9 agonist adjuvant, CpG 1018 at dose of 3000 mcg
  Arms: Z-1018 Dose Level 1
Biological: Z-1018 — contains gE at a dose of 100 mcg to be combined with a Toll-like receptor 9 agonist adjuvant, CpG 1018 at dose of 3000 mcg with aluminum hydroxide (alum)
  Arms: Z-1018 Dose Level 1a
Biological: Z-1018 — contains gE at a dose of 100 mcg to be combined with a Toll-like receptor 9 agonist adjuvant, CpG 1018 at dose of 6000 mcg
  Arms: Z-1018 Dose Level 2
Biological: Z-1018 — contains gE at a dose of 100 mcg to be combined with a Toll-like receptor 9 agonist adjuvant, CpG 1018 at dose of 6000 mcg, with aluminum hydroxide (alum)
  Arms: Z-1018 Dose Level 2a
Biological: Shingrix — a suspension for injection supplied as a single-dose vial of 50 mcg varicella zoster virus (VZV) glycoprotein E (gE) antigen and AS01B adjuvant
  Arms: Shingrix

SUMMARY:
This is a randomized, active-controlled, dose-escalation multi-center study of 2 doses (Day 1 and Week 8) of an investigational herpes zoster (HZ) vaccine (Z-1018), combining herpes zoster antigen- (gE) with a Toll-like receptor 9 (TLR9) agonist adjuvant (CpG 1018) with and without alum in approximately 150 healthy volunteers 50 to 69 years of age (inclusive).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 50 to 69 years of age
* Be in good health in the opinion of the investigator, based upon medical history, physical examination, and laboratory evaluation
* Must be able to comprehend and follow all required study procedures and be available for all visits scheduled in the study
* Seronegative for human immunodeficiency virus (HIV)

Exclusion Criteria:

* History of HZ
* Previous vaccination against varicella or HZ
* If female of childbearing potential, is pregnant, breastfeeding, or planning a pregnancy
* Known history of HIV (HIV 1/2 antibodies)
* Has a history of sensitivity to any component of study vaccines
* Has received any blood products or immunoglobulin within 90 days prior to study injection, or is likely to require infusion of blood products during the study period
* Has received the following prior to the first injection:

  * 14 days: any non-live vaccine
  * 28 days:
  * Any live vaccine, including a COVID-19 vaccine
  * Systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immune suppressive medication, with the exception of inhaled steroids
  * Granulocyte or granulocyte-macrophage colony-stimulating factor
  * Any other investigational medicinal agent, including a COVID-19 vaccine
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose
* Is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of cancer within the last 5 years other than squamous cell or basal cell carcinoma of the skin
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* History of autoimmune disease

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited local and systemic post-injection reactions (PIRs) 7 days after administration of study vaccine | Day 1 to day 7
Frequency of solicited local and systemic post-injection reactions (PIRs) 7 days after administration of study vaccine. | Day 57 to day 63
Number of AEs (Adverse Events) | Day 1 through week 20
Number of SAEs (Serious Adverse Events) | Through week 20

SECONDARY OUTCOMES:
Frequency of CD4+ T cells | At week 12
Measure Geometric mean concentration (GMC) of IgG antibodies to varicella-zoster virus (VZV) antigen glycoprotein E (gE) | At week 12
Response rate of vaccine | At week 12

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Chair — Dynavax Technologies Corporation
Locations (4):
- Australia (4):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Emeritus Research Melbourne, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954